CLINICAL TRIAL: NCT04539951
Title: A Pragmatic Trial of Pharmacotherapy Options Following Unsatisfactory Initial Treatment in OCD
Brief Title: Pragmatic Trial of Obsessive-compulsive Disorder
Acronym: Proceed
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: The first specialized hospital of harbin (Unknown); Guizhou Provincial People's Hospital (Other); First Affiliated Hospital of Jinan University (Other); West China Hospital (Other); Suzhou Psychiatric Hospital (Other); Nanjing Medical University (Other); Wuhan Mental Health Centre (Other); Seventh People's Hospital of Hangzhou (Other); First Affiliated Hospital of Kunming Medical University (Other); General Hospital of Ningxia Medical University (Other); The First Affiliated Hospital of Nanchang University (Other); The Second Affiliated Hospital of Xinxiang Medical University (Unknown)
Responsible Party: Principal Investigator, Zhen Wang, Chief Psychiatrist, Shanghai Mental Health Center
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: CRC2018ZD03
Record Dates: First submitted 2020-08-27; First posted 2020-09-07 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-Compulsive Disorder; Pharmacotherapy; Treatment-naïve; Alternatives
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Fluvoxamine; Venlafaxine Hydrochloride; Memantine; Aripiprazole

STUDY DESIGN:
Intervention Model Description: In phase I all the participants will be initially treated for sertraline for 12 weeks.non-remmitters will be randomly allocated to five treatment arms for another 12 weeks in phase II.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- serotonin treatment (Active Comparator): In experimental phase I, all recruited subjects provide written informed consent before any related procedures. Participants will receive sertraline, initially at 50mg/d, with a weekly 50mg/d further increase, to the maximum recommended dosage (200mg/d) or to the maximum tolerated dosage (less than 200mg/d). Patients will be on their maximum dose by week 4, so allowing an assessment of response at 12 weeks
  Interventions: Drug: Sertraline 200 milligram(mg)
- sequenced treatment alternatives (Active Comparator): If participants in In Experimental phase I do not achieve remission, they will be will be randomly assigned to the second-step treatment (Experimental phase II). The second-step therapy will consist of five treatment options including higher-than-usual-maximal dosage of sertraline, switching to fluvoxamine, switching to venlafaxine, augmentation with memantine, and augmentation with aripiprazole.
  Interventions: Drug: Sertraline 300 milligram(mg); Drug: Fluvoxamine; Drug: Venlafaxine; Drug: Augment with Memantine; Drug: Augment with Aripiprazole

INTERVENTIONS:
Drug: Sertraline 200 milligram(mg) — All included participants will receive sertraline, initially at 50mg/d, with a weekly 50mg/d further increase, to the maximum recommended dosage (200mg/d) or to the maximum tolerated dosage (less than 200mg/d). Patients will be on their maximum dose by week 4, so allowing an assessment of response at 12 weeks
  Arms: serotonin treatment
Drug: Sertraline 300 milligram(mg) — In experimental phase II, the patients in this group will remain on sertraline (higher dosage): where sertraline 200mg has been tolerated, dosage will be increased by 50mg fortnightly to a maximal dose of 300mg/d or to the maximum tolerable dose (less than 300mg/d).
  Arms: sequenced treatment alternatives
Drug: Fluvoxamine — Fluvoxamine will be initiated at a dose of 50mg/d, increasing quickly to a maximal dose of 300mg/d or the maximum tolerated dose by week 4.
  Arms: sequenced treatment alternatives
Drug: Venlafaxine — venlafaxine will be initiated at 75mg/d, increasingly weekly by 75mg/day, to a maximal dose of 300 mg/d or the maximum tolerated dose.
  Arms: sequenced treatment alternatives
Drug: Augment with Memantine — Sertraline will be augmented with memantine initially at 5mg/d, and increasing by 5mg/d weekly to a maximal dose of 20mg/d (10mg twice daily) or the maximum tolerated dose
  Arms: sequenced treatment alternatives
Drug: Augment with Aripiprazole — Sertraline will be augmented with aripiprazole, initially at 5mg/d, and increasing by 5mg/d weekly to a maximal dose of 20mg/d or the maximum tolerated dose
  Arms: sequenced treatment alternatives

SUMMARY:
This study includes a sequenced clinical trial in order to assess the efficacy of several switching or augment strategies when initial treatment is ineffective，and to provide strong evidence for clinical practice and international guidelines for Obsessive-Compulsive Disorder treatments.

DETAILED DESCRIPTION:
Selective Serotonin Reuptake Inhibitors(SSRIs) are the first line pharmacotherapy for Obsessive-Compulsive Disorder (OCD) according to APA（American Psychological Association）guideline. Nevertheless, a large proportion (40% or more) of patients response only partially or not at all to treatment with a SSRI. On the basis of the existing sparse literature, several pharmacotherapy options for OCD patients who do not respond, or who respond but do not remit, have been outlined in current treatment guidelines. These include 1) treatment with higher than usual doses of an SSRI, 2) switch to a different SSRI, 3) switch to a different class of medication, 4) augmentation with a dopamine blocker, and 5) augmentation with a glutamatergic agent. There is a need for additional data, particularly real-world data, on how best to choose between these options.

This proposed Randomized Controlled Trial (RCT) study is a multi-center clinical study with a total of 13 centers that specialize in OCD patients. A randomized block design will be used in this study and all eligible participants accepted into this study will undergo an initial course of pharmacotherapy (phase I), and non-remmitters will be randomly allocated to five treatment arms (phase II). In phase I all participants will be treated with sertraline for 12 weeks.In phase II,The 5 arms will comprise 1) treatment with higher than usual doses of sertraline, 2) switch to fluvoxamine, 3) switch to venlafaxine, 4) augmentation with memantine, and 5) augmentation with aripiprazole. Clinicians and patients will know which treatment arm is being employed, but raters will be kept blind to treatment group.

ELIGIBILITY:
Inclusion criteria:They

* meet DSM-5 diagnostic criteria for OCD as the primary diagnosis ;
* are in the age range from 18 to 65 years;
* have a score of at least 20 on Yale-Brown Obsessive-Compulsive Scale (Y-BOCS);
* have never received medication for OCD, and have not received any form of psychotherapy for OCD in the past 1 month;
* have provided written informed consent.

exclusion criteria: They

* have met the DSM-5 diagnostic criteria for Schizophrenia Spectrum and Other Psychotic Disorders, or the Bipolar and Related Disorders;
* have a moderate or higher risk of suicide (⩾9 on the Suicide Module in the Mini-International Neuropsychiatric Interview (MINI));
* have substance use that is sufficiently severe to possibly impact negatively on treatment adherence in the past 1 year;
* have severe depression with Beck Depression Inventory (BDI) score of ≥29;
* have comorbid psychiatric or medical disorders that may impact negatively on adherence to or on the efficacy of medication (eg borderline personality disorder, CNS disorders)；
* are pregnant or lactating females.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2020-09-22 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) | from baseline to 12 weeks, and 12 weeks to month 6.
  Y-BOCS is a clinician-rated, 10-item scale, each item rated from 0 (no symptoms) to 4 (extreme symptoms), with separate subtotals for severity of obsessions and compulsions.Patients will be assessed at baseline, week 2, week 4, week 8, week 12, week 16, week 20, month 6.

SECONDARY OUTCOMES:
The Clinical Global Impression (CGI) | from 2 weeks to 12 weeks, and 12 weeks to month 6.
  The Clinical Global Impression (CGI; National Institute of Mental Health) is a clinician-rated scale to assess treatment response in patients with mental disorders. The scale contains three items: Severity of Illness; Global Improvement; Efficacy Index. It requires the clinician to rate how much the patient's illness has improved or worsened relative to a baseline measurement. Patients will be assessed at week 2, week 4, week 8, week 12, week 16, week 20, month 6.
Beck Anxiety Inventory (BAI) | from baseline to 12 weeks, and 12 weeks to month 6.
  BAI is a 21-item inventory which identifies anxiety symptoms and quantifies their intensity. Patients will be assessed at baseline, week 2, week 4, week 8, week 12, week 16, week 20, month 6.
Beck Depression Inventory(BDI) | from baseline to 12 weeks, and 12 weeks to month 6.
  BDI is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression.Patients will be assessed at baseline, week 2, week 4, week 8, week 12, week 16, week 20, month 6.
Obsessive-Compulsive Inventory-Revised(OCI-R) | from baseline to 12 weeks, and 12 weeks to month 6.
  OCI-R is the measure of election for the assessment of obsessive-compulsive behaviors, given its validity and the short time that its administration requires. Patients will be assessed at baseline, week 2, week 4, week 8, week 12, week 16, week 20, month 6.
Treatment Emergent Symptom Scale (TESS) | from 2 weeks to 12 weeks , and 12 weeks to month 6.
  The Treatment Emergent Symptom Scale (TESS) is used to record side effects. The side effects are assessed on a five-point scale ranging from 0 ("no side effects") to 4 ("severe side effects"). Patients will be assessed at week 2, week 4, week 8, week 12, week 16, week 20, month 6.
Tolerability scale | from 2 weeks to 12 weeks , and 12 weeks to month 6.
  The tolerability of treatment will be defined as side effect discontinuation in this study. as defined by the proportion of patients who discontinued treatment due to adverse events during the study.Patients will be assessed at week 2, week 4, week 8, week 12, week 16, week 20, month 6.

OTHER OUTCOMES:
Complete Blood Count | baseline
  for safety considerations

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Wang, PhD,MD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang P, Gu W, Gao J, Wang C, Fang J, Hu M, Xiang H, Li B, Liu N, Tang W, Wang X, Jia Y, Li Y, Cheng Y, Tang Z, Simpson HB, Stein DJ, Wang Z. Protocol for a Pragmatic Trial of Pharmacotherapy Options Following Unsatisfactory Initial Treatment in OCD (PROCEED). Front Psychiatry. 2022 May 16;13:822976. doi: 10.3389/fpsyt.2022.822976. eCollection 2022. PMID 35651818